CLINICAL TRIAL: NCT05413265
Title: Alaska Native Family-Based, Financial Incentives Intervention for Smoking Cessation: Phases 1 and 2
Brief Title: Alaska Native Family-Based, Financial Incentives Intervention for Smoking Cessation
Acronym: Aniqsaaq
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Alaska Native Tribal Health Consortium (Other)
Responsible Party: Principal Investigator, Christi Patten, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-000513; 1R01DA056469-01A1 (NIH)
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Smoking Cessation
Keywords: Alaska Native; Smoking Cessation; Family; Financial Incentive
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phases 1 and 2 (Other): Phase 1 participants will help inform the cultural adaptation of the study design and materials. Phase 2 will enroll 10 dyads (20 individuals) of AN/AI people who smoke and a family member. Dyad participants will help beta-test the feasibility and acceptability of the financial incentives intervention.
  Interventions: Behavioral: Phases 1 and 2

INTERVENTIONS:
Behavioral: Phases 1 and 2 — Phase 1 participants will help inform the cultural adaptation of the study design and materials. Phase 2 will enroll 10 dyads (20 individuals) of AN/AI people who smoke and a family member. Dyad participants will help beta-test the feasibility and acceptability of the financial incentives intervention.

SUMMARY:
The objective of the proposed study is to develop and beta-test a culturally adapted, Alaska Native family-based incentives intervention for smoking cessation.

DETAILED DESCRIPTION:
Aim 1 has two phases:

In Aim 1/Phase 1, we will use qualitative in-depth individual interviews to culturally tailor and adapt the intervention. These interviews (n=36) will include Alaska Native or American Indian (AN/AI) people who smoke (n=12), family members of Alaska Native people who smoke (n=12), and stakeholders from the Alaska Tribal Health System (n=12). We will present the proposed financial incentives intervention to each group and ask them questions about possible concerns, recruitment strategies, possible risks, and appeal to Alaska Native culture. For the stakeholders, we will also ask about potential barriers of implementing the program into their organization/department.

In Aim 1/Phase 2, we will beta-test and refine the intervention with 10 dyads comprising of an AN/AI person who smokes and their family member. The beta-test will last for 6 months. The dyad will receive cash rewards of increasing value over the course of the 6 months for negative, completed smoking status checks. A negative check-in counts as self-reported abstinence and biochemically confirmed abstinence: saliva cotinine sample measuring ≤ 30 n/ml (negative Alere iScreen result) and expired carbon monoxide sample measuring ≤ 6 ppm with iCOQuit device.

ELIGIBILITY:
Inclusion Criteria:

Index Participants will be eligible if they:

* Are an ANAI person (based on self-reported race/ethnicity) and reside in Alaska.
* Are aged ≥ 18 years (legal smoking age in Alaska).
* Self-report smoking in the past 7 days, biochemically verified with saliva cotinine ≥ 30 n/ml (positive Alere iScreen result) for Phase 2.
* Smoked ≥ 3 cigarettes per day (cpd) over the past 3 months.
* If other tobacco or nicotine product used, cigarettes are the main tobacco product used.
* Are considering or willing to make a quit attempt.
* Own or have access to a mobile phone or tablet with Internet and text messaging capabilities, or will be loaned an iPad mini for the study duration.
* Nominate one adult family member who will enroll.

Index Participants Exclusion Criteria:

* Used pharmacotherapy or a stop smoking program within the past 3 months.
* Another person in the household is enrolled as the index participant.
* Smokes marijuana at least once a week and not willing to quit for study (interferes with breath test) in Phase 2

Family Member Participants, regardless of smoking status or residence with the index participant, will be eligible if they:

* Are ≥ 18 years old.
* Are defined as family by the index participant.
* Own or have access to a mobile phone or tablet with internet and text messaging capabilities or will be loaned an iPad mini for the study duration.
* Both men and women and those from non-ANAI racial/ethnic groups.
* Family members may only support one index participant.

Alaska Tribal Health System stakeholders (Phase 1 only):

- Input from healthcare providers, cessation specialists, and THO leaders will be gathered to understand potential facilitators and barriers to adoption of the intervention within the ATHS. The ANTHC team will invite individuals to participate through phone and email communications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Change in smoking status | 6 months, 12 months
  Number of participants to have biochemically confirmed, prolonged smoking abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Christi A Patten, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Patten CA, Koller KR, King DK, Prochaska JJ, Sinicrope PS, McDonell MG, Decker PA, Lee FR, Fosi JK, Young AM, Sabaque CV, Brown AR, Borah BJ, Thomas TK. Aniqsaaq (To Breathe): Study protocol to develop and evaluate an Alaska Native family-based financial incentive intervention for smoking cessation. Contemp Clin Trials Commun. 2023 Apr 3;33:101129. doi: 10.1016/j.conctc.2023.101129. eCollection 2023 Jun. PMID 37091507
- [Result] Sinicrope PS, Tranby BN, Young AM, Koller KR, King DK, Lee FR, Sabaque CV, Prochaska JJ, Borah BJ, Decker PA, McDonell MG, Stillwater B, Thomas TK, Patten CA. Adapting a Financial Incentives Intervention for Smoking Cessation With Alaska Native Families: Phase 1 Qualitative Research to Inform the Aniqsaaq (To Breathe) Study. Nicotine Tob Res. 2024 Sep 23;26(10):1377-1384. doi: 10.1093/ntr/ntae092. PMID 38642396
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20539920

DOCUMENTS (1):
  • Informed Consent Form (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT05413265/ICF_000.pdf